CLINICAL TRIAL: NCT02635204
Title: A Randomized, Double-Blind, Vehicle-Controlled, Multicenter, Parallel Group Study of the Efficacy and Safety of DFD-06 Cream in the Treatment of Moderate to Severe Plaque Psoriasis for 14 Days
Brief Title: A Study of the Efficacy and Safety of DFD-06 Cream in the Treatment of Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Promius Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFD06-CD-004
Record Dates: First submitted 2015-12-08; First posted 2015-12-18 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DFD-06 Cream (Experimental): DFD-06 Cream will be applied to subjects with moderate plaque psoriasis twice daily for 14 days.
  Interventions: Drug: DFD06 Cream
- Vehicle Cream (Placebo Comparator): Vehicle Cream will be applied to subjects with moderate plaque psoriasis twice daily for 14 days.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: DFD06 Cream — Twice daily topical application for 14 days.
  Other Names: Clobetasol propionate Cream, 0.025%
  Arms: DFD-06 Cream
Drug: Vehicle Cream — Twice daily topical application for 14 days.
  Arms: Vehicle Cream

SUMMARY:
This study will compare the efficacy and safety of DFD-06 Cream to Vehicle Cream for topical treatment of moderate to severe plaque psoriasis after 3, 7, and 14 days of treatment.

DETAILED DESCRIPTION:
This study will be a multicenter (approximately 30 sites), randomized, vehicle-controlled, double-blind, and parallel group design. Approximately 264 subjects with moderate to severe plaque psoriasis will be randomized to treatment with DFD-06 Cream or Vehicle Cream. Subjects will use study product twice daily for 14 days. Subject visits are scheduled at Screening, Baseline (Day 1) and Days 4, 8, and 15. Clinical determinations of disease severity will be performed using the total sign score (TSS) for the target lesion and Investigator Global Assessment (IGA) for overall severity.

ELIGIBILITY:
Inclusion Criteria:

1. Subject understands the study procedures and agrees to participate by giving written informed consent. Subjects must be willing to authorize use and disclosure of protected health information collected for the study.
2. Subject must be at least 18 years of age.
3. Subject must present with a clinical diagnosis of stable (at least 3 months) plaque-type psoriasis.
4. Subject with psoriasis involving 3% or greater BSA, not including the face, scalp, groin, axillae and other intertriginous areas.
5. Subject must have an IGA grade of 3 or 4 (moderate to severe) at the Baseline Visit.
6. Female subjects of childbearing potential must agree to use contraception during the study which can include abstinence with an adequate secondary option should the subject become sexually active. All women of childbearing potential must complete a urine pregnancy test (test must have a sensitivity of at least 25mIU/ml for human chorionic gonadotropin) at the Baseline Visit (Visit 2) and the test result must be negative to be eligible for enrollment.
7. Subject must be in good general health as determined by the investigator and supported by the medical history and normal or not clinically significant abnormal vital signs (blood pressure and pulse).

Exclusion Criteria:

1. Current diagnosis of unstable forms of psoriasis including guttate, erythrodermic, exfoliative or pustular psoriasis.
2. Other inflammatory skin disease that may confound the evaluation of the plaque psoriasis (e.g., atopic dermatitis, contact dermatitis, tinea corporis).
3. Presence of pigmentation, extensive scarring, or pigmented lesions or sunburn which could interfere with the rating of efficacy parameters.
4. History of psoriasis unresponsive to biological or topical treatments.
5. History of organ transplant requiring immunosuppression, HIV, or other immunocompromised state.
6. Use within 180 days prior to Baseline Visit of biologic treatment for psoriasis (e.g., infliximab, adalimumab, etanercept, ustekinumab, secukinumab, or alefacept).
7. Have received treatment for any type of cancer within 5 years of the Baseline Visit except skin cancer and cervical cancer (in situ) are allowed if at least 1 year before the Baseline Visit.
8. Use within 60 days prior to the Baseline Visit of: 1) systemic or topical immunosuppressive drugs (e.g., tacrolimus, pimecrolimus), 2) systemic antipsoriatic treatment (e.g., methotrexate, cyclosporine, hydroxyurea) or 3) oral retinoids (e.g., acitretin, isotretinoin).
9. Use within 30 days prior to the Baseline Visit of: 1) systemic steroids, 2) PUVA therapy, 3) systemic anti-inflammatory agents (e.g., mycophenolate mofetil, sulfasalazine, 6-thioguanine), or 4) UVB therapy. Inhaled, intraocular, and intranasal steroids are allowed.
10. Use within 14 days prior to the Baseline Visit of: 1) topical antipsoriatic drugs (e.g., salicylic acid, anthralin, coal tar, calcipotriene), 2) topical retinoids (e.g., tazarotene, tretinoin) or 3) topical corticosteroids.
11. Subjects who have participated in a study of an investigational drug 60 days prior to the Baseline Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Sidgiddi, MD, Study Director — Dr. Reddy's Laboratories, Inc
Locations (30):
- United States (30):
  - Site 116, Glendale, Arizona
  - Site 111, Rogers, Arkansas
  - Site 124, Fountain Valley, California
  - Site 120, Laguna Hills, California
  - Site 122, San Diego, California
  - Site 123, San Diego, California
  - Site 113, Denver, Colorado
  - Site 117, New Haven, Connecticut
  - Site 108, Brandon, Florida
  - Site 112, Coral Gables, Florida
  - Site 106, Jacksonville, Florida
  - Site 110, Pinellas Park, Florida
  - 130, West Palm Beach, Florida
  - Site 103, Arlington Heights, Illinois
  - Site 115, Overland Park, Kansas
  - Site 127, Beverly, Massachusetts
  - Site 119, Quincy, Massachusetts
  - 129, Henderson, Nevada
  - Site 114, New York, New York
  - Site 104, Rocky Mount, North Carolina
  - Site 105, Wilmington, North Carolina
  - Site 126, Cincinnati, Ohio
  - Site 121, Warwick, Rhode Island
  - Site 107, Nashville, Tennessee
  - 128, Arlington, Texas
  - Site 101, Dallas, Texas
  - Site 102, Houston, Texas
  - Site 109, San Antonio, Texas
  - Site 118, Norfolk, Virginia
  - Site 125, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DFD-06 Cream: DFD-06 Cream was applied to subjects with moderate plaque psoriasis twice daily for 14 days.
- Vehicle Cream: Vehicle Cream was applied to subjects with moderate plaque psoriasis twice daily for 14 days.
Period: Overall Study
Arm/Group | DFD-06 Cream | Vehicle Cream
Started | 178 | 89
Completed | 176 | 88
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- DFD-06 Cream: Participants applied DFD-06 Cream twice daily for 14 days.
- Vehicle Cream: Participants received Vehicle Cream and was applied twice daily for 14 days.
- Total: Total of all reporting groups
Arm/Group | DFD-06 Cream | Vehicle Cream | Total
Number analyzed (Participants) | 178 | 89 | 267
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 151 | 75 | 226
  >=65 years | 27 | 14 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (13.59) | 50.6 (15.93) | 49.8 (14.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 45 | 123
  Male | 100 | 44 | 144
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 178 | 89 | 267

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Treatment Success at Day 15
Description: The percentage of subjects with treatment success (defined as IGA = 0 or 1 and at least a 2-grade reduction from baseline) at the Day 15 visit. Primary analysis was done with multiple imputations. Results are combined analyses from 5 imputed data sets.
Time Frame: Day 15 Visit
Population: Intention to treat population defined as all subjects who were randomized and dispensed medication
Measure: Number; unit: percentage of participants
Groups:
- DFD-06 Cream: Participants received DFD-06 Cream applied topical twice daily for 14 days.
- Vehicle Cream: Participants received Vehicle Cream applied topical twice daily for 14 days.
Arm/Group | DFD-06 Cream | Vehicle Cream
Number analyzed (Participants) | 178 | 89
percentage of participants | 30.2 | 9.0

2. Secondary Outcome: Percent Change From Baseline in Body Surface Area at Day 15
Description: Percent change from baseline in body surface area affected by psoriasis at Day 15. The analysis was done with multiple imputations. Results are combined analyses from 5 imputed data sets.
Time Frame: Baseline and Day 15
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: percentage change in body surface area
Arm/Group | DFD-06 Cream | Vehicle Cream
Number analyzed (Participants) | 178 | 89
percentage change in body surface area | -28.9 (34.00) | -6.1 (32.67)

3. Secondary Outcome: Percent of Subjects With Treatment Success at Day 8 Visit
Description: Percent of subjects with treatment success at Day 8 Visit defined as an IGA of 0 or 1 with at least a 2 grade reduction from baseline. The analysis was done with multiple imputations. Results are combined analyses from 5 imputed data sets.
Time Frame: Baseline and Day 8
Population: Intention to treat population defined as all subjects who were randomized and dispensed medication
Measure: Number; unit: percentage of subject
Arm/Group | DFD-06 Cream | Vehicle Cream
Number analyzed (Participants) | 178 | 89
percentage of subject | 15.7 | 5.6

ADVERSE EVENTS:
Time Frame: Baseline to Day 15 Visit
Description: Subjects queried at every visit for Adverse Events
Groups:
- DFD-06 Cream: DFD-06 Cream applied to subjects twice daily for 14 days.
- Vehicle Cream: Vehicle Cream applied to subjects twice daily for 14 days.
Arm/Group | DFD-06 Cream | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/178 | 0/89
Serious Adverse Events (participants affected / at risk) | 1/178 | 0/89
Other Adverse Events (participants affected / at risk) | 24/178 | 17/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFD-06 Cream (N=178) | Vehicle Cream (N=89)
Metastatic Lymphoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFD-06 Cream (N=178) | Vehicle Cream (N=89)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
application site discolouration (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Application Site Fissure (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Application Site Pain (Skin and subcutaneous tissue disorders) | 8 (8) | 7 (7)
Application Site Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 8 (8)
Application site Telangiectasia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infections and Infestations (Infections and infestations) | 2 (2) | 0 (0)
Application site Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cronic hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Nervous System Disorders (Nervous system disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cirrhosis Alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No